CLINICAL TRIAL: NCT00394277
Title: Randomized, Multicenter, Double-blinded, Phase IV Study Evaluating the Efficacy (as Measured by Sustained Virological Response) and Safety of 360 μg Induction Dosing of Pegasys® in Combination With Higher Copegus® Doses in Treatment-naïve Patients With Chronic Hepatitis C Genotype 1 Virus Infection of High Viral Titer and Baseline Body Weight Greater Than or Equal to 85 kg
Brief Title: A Study of Induction Dosing With PEGASYS (Peginterferon Alfa-2a [40KD]) Plus Copegus in Treatment-Naive Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NV18210
Record Dates: First submitted 2006-10-30; First posted 2006-10-31 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- PEG-IFN 180 µg + Ribavirin 1200 mg (Experimental)
  Interventions: Drug: peginterferon alfa-2a; Drug: Ribavirin
- PEG-IFN 180 µg + Ribavirin 1400/1600 mg (Experimental)
  Interventions: Drug: peginterferon alfa-2a; Drug: Ribavirin
- PEG-IFN 360/180 µg + Ribavirin 1200 mg (Experimental)
  Interventions: Drug: Ribavirin; Drug: peginterferon alfa-2a
- PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg (Experimental)
  Interventions: Drug: peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: peginterferon alfa-2a — 180 µg sc weekly for 48 weeks
  Other Names: Pegasys
  Arms: PEG-IFN 180 µg + Ribavirin 1200 mg; PEG-IFN 180 µg + Ribavirin 1400/1600 mg
Drug: Ribavirin — 1200 mg po daily for 48 weeks
  Other Names: Copegus
  Arms: PEG-IFN 180 µg + Ribavirin 1200 mg; PEG-IFN 360/180 µg + Ribavirin 1200 mg
Drug: peginterferon alfa-2a — 360 µg sc weekly decreasing to 180 µg sc weekly for 48 weeks
  Other Names: Pegasys
  Arms: PEG-IFN 360/180 µg + Ribavirin 1200 mg; PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg
Drug: Ribavirin — 1400-1600 mg po daily for 48 weeks
  Other Names: Copegus
  Arms: PEG-IFN 180 µg + Ribavirin 1400/1600 mg; PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg

SUMMARY:
This 4-arm study will compare the efficacy and safety of PEGASYS induction and maintenance dosing, versus standard fixed dosing in combination with Copegus, and the efficacy and safety of higher dose versus standard dose Copegus in combination with PEGASYS. Patients with chronic hepatitis C (CHC) genotype 1 infection of high viral titer, and baseline body weight ≥85 kg, will be randomized to one of 4 groups, to receive one of the following: a) PEGASYS 180 µg subcutaneously (sc) weekly plus Copegus 1200 mg orally (po) daily; b) PEGASYS 180 µg sc weekly plus Copegus 1400-1600 mg po daily; c)PEGASYS 360 µg sc weekly (induction) followed by 180 µg sc weekly (maintenance) plus Copegus 1200 mg po daily; or d) PEGASYS 360 µg sc weekly (induction) followed by 180 µg sc weekly (maintenance) plus Copegus 1400-1600 mg po daily. Following 48 weeks treatment, there will be a 24-week period of treatment-free follow-up. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥18 years of age
* CHC infection, genotype 1
* Hepatitis C virus (HCV) RNA ≥400,000 IU/mL
* Baseline body weight ≥85 kg
* Liver biopsy (within 24 months of first dose) with results consistent with CHC

Exclusion Criteria:

* Previous treatment with interferon, ribavirin, viramidine, levovirin, HCV polymerase or protease inhibitors
* Other forms of liver disease, including liver cancer
* Human immunodeficiency virus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1175 (Actual)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (152):
- United States (77):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Fresno, California
  - La Jolla, California
  - Lancaster, California
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - San Luis Obispo, California
  - San Marcos, California
  - Ventura, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Sarasota, Florida
  - Atlanta, Georgia
  - Austell, Georgia
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Winfield, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Ypsilanti, Michigan
  - Plymouth, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Egg Harbour Township, New Jersey
  - Vineland, New Jersey
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Williamsville, New York
  - Yonkers, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Fayetteville, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Cranston, Rhode Island
  - Providence, Rhode Island
  - Columbia, South Carolina
  - Germantown, Tennessee
  - West Nashville, Tennessee
  - Dallas, Texas
  - Fort Sam Houston, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Annandale, Virginia
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Fairfax, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Tacoma, Washington
  - Vancouver, Washington
  - Casper, Wyoming
  - Cheyenne, Wyoming
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Brazil (7):
  - Caixa
  - Campinas
  - Juiz de Fora
  - Porto Alegre
  - Salvador
  - São José do Rio Preto
  - São Paulo
- Canada (8):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Denmark (2):
  - Kolding
  - Odense
- France (6):
  - Clermont-Ferrand
  - Clichy
  - Lille
  - Lyon
  - Rouen
  - Strasbourg
- Germany (12):
  - Berlin
  - Bonn
  - Cologne
  - Düsseldorf
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Giessen
  - Hamburg
  - Hanover
  - Heidelberg
  - Kiel
  - Tübingen
- Hungary (7):
  - Békéscsaba
  - Budapest
  - Debrecen
  - Győr
  - Gyula
  - Pécs
  - Szombathely
- Netherlands (3):
  - Amsterdam
  - Leiden
  - Rotterdam
- Poland (6):
  - Bydgoszcz
  - Chorzów
  - Kielce
  - Lodz
  - Warsaw
  - Wroclaw
- Puerto Rico (3):
  - Ponce
  - San Juan
  - Santurce
- Romania (5):
  - Bucharest
  - Cluj-Napoca
  - Constanța
  - Iași
  - Timișoara
- Russia (7):
  - Jaloslave
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Samara
  - Smolensk
  - Stavropol
- Sweden (2):
  - Stockholm
  - Uppsala
- United Kingdom (4):
  - London
  - Newcastle upon Tyne
  - Plymouth
  - Southampton

REFERENCES:
- [Derived] Reddy KR, Shiffman ML, Rodriguez-Torres M, Cheinquer H, Abdurakhmanov D, Bakulin I, Morozov V, Silva GF, Geyvandova N, Stanciu C, Rabbia M, McKenna M, Thommes JA, Harrison SA; PROGRESS Study Investigators. Induction pegylated interferon alfa-2a and high dose ribavirin do not increase SVR in heavy patients with HCV genotype 1 and high viral loads. Gastroenterology. 2010 Dec;139(6):1972-83. doi: 10.1053/j.gastro.2010.08.051. Epub 2010 Sep 30. PMID 20816836

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG-IFN 180 µg + Ribavirin 1200 mg: PEG-IFN 180 µg administered subcutaneously once weekly in abdomen or thigh. Ribavirin 600 mg administered orally twice daily (total of 1200 mg daily).
- PEG-IFN 180 µg + Ribavirin 1400/1600 mg: PEG-IFN 180 µg administered subcutaneously once weekly in abdomen or thigh. Patients with a body weight of 85 kg to <95 kg took 600 mg of ribavirin (3 tablets) in the morning and 800 mg (4 tablets) in the evening, or vice versa; total daily dose was 1400 mg. Patients with a body weight ≥ 95 kg took 800 mg of ribavirin (4 tablets) in the morning and evening; total daily dose was 1600 mg.
- PEG-IFN 360/180 µg + Ribavirin 1200 mg: PEG-IFN 360 or 180 µg administered subcutaneously once weekly in abdomen or thigh. Ribavirin 600 mg administered orally twice daily (total of 1200 mg daily).
- PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg: PEG-IFN 360 or 180 µg administered subcutaneously once weekly in abdomen or thigh. Patients with a body weight of 85 kg to <95 kg took 600 mg of ribavirin (3 tablets) in the morning and 800 mg (4 tablets) in the evening, or vice versa; total daily dose was 1400 mg. Patients with a body weight ≥ 95 kg took 800 mg of ribavirin (4 tablets) in the morning and evening; total daily dose was 1600 mg.
Period: Overall Study
Arm/Group | PEG-IFN 180 µg + Ribavirin 1200 mg | PEG-IFN 180 µg + Ribavirin 1400/1600 mg | PEG-IFN 360/180 µg + Ribavirin 1200 mg | PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg
Started | 195 | 196 | 393 | 391
Completed | 137 | 136 | 273 | 266
Not Completed | 58 | 60 | 120 | 125

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG-IFN 180 µg + Ribavirin 1200 mg | PEG-IFN 180 µg + Ribavirin 1400/1600 mg | PEG-IFN 360/180 µg + Ribavirin 1200 mg | PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg | Total
Number analyzed (Participants) | 195 | 196 | 393 | 391 | 1175
Age Continuous [Mean (Standard Deviation); unit: years] — Intent-to-treat population (all patients treated with at least one dose of either study medication) PEG-IFN 180 µg + Ribavirin 1200 mg: n = 191 PEG-IFN 180 µg + Ribavirin 1400/1600 mg: n = 189 PEG-IFN 360/180 µg + Ribavirin 1200 mg: n = 382 PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg: n = 383
  years | 46.1 (9.86) | 45.1 (9.50) | 45.7 (9.64) | 46.0 (10.18) | 45.7 (9.83)
Gender [Number; unit: Patients] — Intent-to-treat population (all patients treated with at least one dose of either study medication) PEG-IFN 180 µg + Ribavirin 1200 mg: n = 191 PEG-IFN 180 µg + Ribavirin 1400/1600 mg: n = 189 PEG-IFN 360/180 µg + Ribavirin 1200 mg: n = 382 PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg: n = 383
  Patients
    Female | 37 | 41 | 90 | 73 | 241
    Male | 154 | 148 | 292 | 310 | 904

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response (SVR)-24 (Scheduled Treatment Period)
Description: SVR-24 according to the scheduled treatment period was defined as the percentage of patients with undetectable HCV RNA at 24 weeks after completion of the treatment period (a single last HCV RNA PCR <15 IU/mL measured at or after week 68 (ie, on or after study day 477).
Time Frame: Week 72
Population: Intent-to-treat population (all patients treated with at least one dose of either study medication)
Measure: Number; unit: Percentage of patients
Arm/Group | PEG-IFN 180 µg + Ribavirin 1200 mg | PEG-IFN 180 µg + Ribavirin 1400/1600 mg | PEG-IFN 360/180 µg + Ribavirin 1200 mg | PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg
Number analyzed (Participants) | 191 | 189 | 382 | 383
Percentage of patients | 37.7 | 42.9 | 43.5 | 40.7
Statistical Analysis 1: Comparison: PEG-IFN 180 µg + Ribavirin 1200 mg vs PEG-IFN 180 µg + Ribavirin 1400/1600 mg vs PEG-IFN 360/180 µg + Ribavirin 1200 mg vs PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg; This reflects the primary protocol-specified comparison (standard Pegasys induction dosing arms versus pooled Pegasys induction dosing arms). The study was designed to have at least 86% power for testing the null hypothesis of no difference between these two pooled groups, with assumed response rates of 28%, 32%, 36%, and 43% in the four treatment arms; Test type: Superiority or Other; p = 0.584, Cochran-Mantel-Haenszel — All secondary comparisons were tested at a two-sided significance level of 0.05; P-value obtained from CMH test, stratified by country and ribavirin dose strata; Odds Ratio (OR) = 1.075, 95% CI [0.831 to 1.391]

2. Secondary Outcome: SVR-24 (Actual Treatment Period)
Description: SVR-24 according to the actual treatment period was defined as the percentage of patients with undetectable HCV RNA at least 20 weeks after the last dose of study drug.
Time Frame: 24 weeks after end of treatment
Population: Intent-to-treat population (all patients treated with at least one dose of either study medication)
Measure: Number; unit: Percentage of patients
Arm/Group | PEG-IFN 180 µg + Ribavirin 1200 mg | PEG-IFN 180 µg + Ribavirin 1400/1600 mg | PEG-IFN 360/180 µg + Ribavirin 1200 mg | PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg
Number analyzed (Participants) | 191 | 189 | 382 | 383
Percentage of patients | 38.2 | 43.9 | 43.5 | 40.7
Statistical Analysis 1: Comparison: PEG-IFN 180 µg + Ribavirin 1200 mg vs PEG-IFN 180 µg + Ribavirin 1400/1600 mg vs PEG-IFN 360/180 µg + Ribavirin 1200 mg vs PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg; (PEG-IFN 180 µg + Ribavirin 1200 mg and PEG-IFN 180 µg + Ribavirin 1400/1600 mg) vs. (PEG-IFN 360/180 µg + Ribavirin 1200 mg and PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg); Test type: Superiority or Other; p = 0.775, Cochran-Mantel-Haenszel — All secondary comparisons are tested at a two-sided significance level of 0.05; P-value obtained from CMH test, stratified by country and ribavirin dose strata; Odds Ratio (OR) = 1.039, 95% CI [0.803 to 1.344]

3. Secondary Outcome: SVR-12 (Scheduled Treatment Period)
Description: SVR-12 according to the scheduled treatment period was defined as the percentage of patients with undetectable HCV RNA at 12 weeks after the scheduled treatment period (a single last HCV RNA PCR <15 IU/mL measured at or after week 60).
Time Frame: 12 weeks after end of treatment
Population: Intent-to-treat population (all patients treated with at least one dose of either study medication)
Measure: Number; unit: Percentage of patients
Arm/Group | PEG-IFN 180 µg + Ribavirin 1200 mg | PEG-IFN 180 µg + Ribavirin 1400/1600 mg | PEG-IFN 360/180 µg + Ribavirin 1200 mg | PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg
Number analyzed (Participants) | 191 | 189 | 382 | 383
Percentage of patients | 40.3 | 45.0 | 44.2 | 41.5
Statistical Analysis 1: Comparison: PEG-IFN 180 µg + Ribavirin 1200 mg vs PEG-IFN 180 µg + Ribavirin 1400/1600 mg vs PEG-IFN 360/180 µg + Ribavirin 1200 mg vs PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.973, Cochran-Mantel-Haenszel — All secondary comparisons are tested at a two-sided significance level of 0.05; P-value obtained from CMH test, stratified by country and ribavirin dose strata; Odds Ratio (OR) = 1.004, 95% CI [0.777 to 1.299]

4. Secondary Outcome: SVR-12 (Actual Treatment Period)
Description: SVR-12 according to the actual treatment period was defined as the percentage of patients with undetectable HCV RNA at least 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after end of treatment
Population: Intent-to-treat population (all patients treated with at least one dose of either study medication)
Measure: Number; unit: Percentage of patients
Arm/Group | PEG-IFN 180 µg + Ribavirin 1200 mg | PEG-IFN 180 µg + Ribavirin 1400/1600 mg | PEG-IFN 360/180 µg + Ribavirin 1200 mg | PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg
Number analyzed (Participants) | 191 | 189 | 382 | 383
Percentage of patients | 40.3 | 45.5 | 44.2 | 42.3
Statistical Analysis 1: Comparison: PEG-IFN 180 µg + Ribavirin 1200 mg vs PEG-IFN 180 µg + Ribavirin 1400/1600 mg vs PEG-IFN 360/180 µg + Ribavirin 1200 mg vs PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.951, Cochran-Mantel-Haenszel — All secondary comparisons are tested at a two-sided significance level of 0.05; P-value obtained from CMH test, stratified by country and ribavirin dose strata; Odds Ratio (OR) = 1.008, 95% CI [0.780 to 1.304]

ADVERSE EVENTS:
Arm/Group | PEG-IFN 180 µg + Ribavirin 1200 mg | PEG-IFN 180 µg + Ribavirin 1400/1600 mg | PEG-IFN 360/180 µg + Ribavirin 1200 mg | PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg
Serious Adverse Events (participants affected / at risk) | 22/191 | 20/189 | 36/382 | 39/383
Other Adverse Events (participants affected / at risk) | 186/191 | 179/189 | 370/382 | 373/383
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN 180 µg + Ribavirin 1200 mg (N=191) | PEG-IFN 180 µg + Ribavirin 1400/1600 mg (N=189) | PEG-IFN 360/180 µg + Ribavirin 1200 mg (N=382) | PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg (N=383)
Pneumonia (Infections and infestations) | 1 | 3 | 2 | 4
Appendicitis (Infections and infestations) | 0 | 0 | 3 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 2 | 0
Abscess Limb (Infections and infestations) | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 2 | 0 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Bursitis Infective (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0 | 0
Injection Site Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Intervertebral Discitis (Infections and infestations) | 0 | 0 | 1 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Lung Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Pelvic Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pelvic Inflammatory Disease (Infections and infestations) | 0 | 0 | 1 | 0
Rectal Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 3 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 2 | 0
Acute Psychosis (Psychiatric disorders) | 0 | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Completed Suicide (Psychiatric disorders) | 0 | 0 | 1 | 0
Dependence (Psychiatric disorders) | 1 | 0 | 0 | 0
Hostility (Psychiatric disorders) | 0 | 0 | 1 | 0
Major Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Panic Attack (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Anaemia Haemolytic Autoimmune (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1
Altered State of Consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Metabolic Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 2
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Postoperative Fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Venom Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Gait Disturbance (General disorders) | 0 | 0 | 1 | 0
Hyperplasia (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0
Multi-Organ Failure (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatorenal Syndrome (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Retinal Haemorrhage (Eye disorders) | 1 | 1 | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 1 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Alveolitis Fibrosing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fracture Nonunion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 0 | 0 | 2 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Tubulointerstitial Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Vena Cava Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN 180 µg + Ribavirin 1200 mg (N=191) | PEG-IFN 180 µg + Ribavirin 1400/1600 mg (N=189) | PEG-IFN 360/180 µg + Ribavirin 1200 mg (N=382) | PEG-IFN 360/180 µg + Ribavirin 1400/1600 mg (N=383)
Pyrexia (General disorders) | 83 | 78 | 176 | 205
Fatigue (General disorders) | 66 | 102 | 184 | 182
Chills (General disorders) | 42 | 55 | 122 | 132
Asthenia (General disorders) | 28 | 35 | 84 | 80
Irritability (General disorders) | 34 | 29 | 64 | 66
Pain (General disorders) | 10 | 18 | 24 | 31
Injection Site Erythema (General disorders) | 16 | 14 | 28 | 24
Injection Site Reaction (General disorders) | 12 | 13 | 20 | 14
Malaise (General disorders) | 10 | 10 | 14 | 18
Nausea (Gastrointestinal disorders) | 41 | 42 | 112 | 104
Diarrhoea (Gastrointestinal disorders) | 25 | 27 | 62 | 62
Vomiting (Gastrointestinal disorders) | 12 | 19 | 42 | 31
Abdominal Pain Upper (Gastrointestinal disorders) | 11 | 18 | 28 | 23
Dyspepsia (Gastrointestinal disorders) | 9 | 12 | 25 | 23
Dry Mouth (Gastrointestinal disorders) | 5 | 14 | 23 | 23
Abdominal Pain (Gastrointestinal disorders) | 6 | 10 | 15 | 13
Constipation (Gastrointestinal disorders) | 5 | 13 | 9 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 46 | 44 | 111 | 118
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 | 49 | 88 | 89
Back Pain (Musculoskeletal and connective tissue disorders) | 21 | 22 | 28 | 23
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 8 | 12 | 13 | 15
Rash (Skin and subcutaneous tissue disorders) | 38 | 40 | 65 | 78
Pruritus (Skin and subcutaneous tissue disorders) | 34 | 27 | 76 | 59
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 20 | 71 | 71
Dry Skin (Skin and subcutaneous tissue disorders) | 23 | 22 | 38 | 37
Headache (Nervous system disorders) | 75 | 76 | 151 | 168
Dizziness (Nervous system disorders) | 14 | 27 | 44 | 59
Disturbance in Attention (Nervous system disorders) | 5 | 6 | 20 | 27
Insomnia (Psychiatric disorders) | 46 | 45 | 98 | 113
Depression (Psychiatric disorders) | 31 | 33 | 65 | 56
Anxiety (Psychiatric disorders) | 11 | 18 | 31 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 35 | 59 | 69
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 15 | 39 | 32
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 16 | 22
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 13 | 17 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 9 | 14
Anaemia (Blood and lymphatic system disorders) | 23 | 22 | 38 | 54
Neutropenia (Blood and lymphatic system disorders) | 9 | 16 | 29 | 28
Decreased Appetite (Metabolism and nutrition disorders) | 30 | 31 | 73 | 85
Weight Decreased (Investigations) | 31 | 31 | 54 | 67
Hypertension (Vascular disorders) | 7 | 11 | 16 | 20
Upper Respiratory Tract Infection (Infections and infestations) | 11 | 7 | 11 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.